CLINICAL TRIAL: NCT00225628
Title: Improving Quality With Outpatient Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5U18HS011046 (AHRQ)
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2005-09-26 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease; Osteoporosis; Hypertension; Hyperlipidemia
Keywords: Computerized clinical decision support; Patient Safety; Quality of Care; Electronic Medical Records; Chronic Disease Management; Drug Monitoring; Guideline Adherence; Reminder Systems
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Osteoporosis; Hypertension; Hyperlipidemias

INTERVENTIONS:
Behavioral: Computerized Reminders Medications Monitoring
Behavioral: Computerized Test Results Management Application
Behavioral: Computerized Reminders Hypertension Management
Behavioral: Computerized Reminders Osteoporosis Screening and Mgt

SUMMARY:
Assesses physician compliance with paper-based and electronic guidelines, reminders, and alerts for outpatient settings. Target areas for the reminders and alerts are disease management, medication management, and interpretation of abnormal test results.

DETAILED DESCRIPTION:
The evidence base for practicing medicine continues to improve. However, abundant data show that gaps exist between best evidence and practice. Moreover, health care costs are climbing at an alarming rate. We propose to ask three related questions: 1) how effective are computer decision-support systems for improving compliance with evidence-based guidelines and costs in the ambulatory setting; 2) what is the impact on guideline compliance of applications that allow clinicians to track and follow-up test results; and 3) what are the main barriers to acceptance of guidelines delivered via real-time clinical decision-support systems.

Our work and that of others has shown that computerized decision-support in the form of alerts and reminders can improve outcomes and reduce costs in the inpatient setting. However, fewer data are available in the outpatient setting. An elegant series of studies from Regenstrief found that certain computer-based interventions, such as displaying charges for tests, prior test results, and the likelihood that a particular test would be abnormal, all reduced outpatient utilization, and that reminders to perform health maintenance procedures improved compliance. However, such systems are still not used broadly and the full potential of computer-based technology remains to be tested.

Also, there is ample evidence that physicians do not always act optimally on the results of patient studies and often are remiss at communicating satisfactorily with patients about the results of these studies. This situation may be exacerbated by increasing patient volumes in the face of managed care. The ability of the computer to assist in the tracking and follow-up of test results as well as communication with patients remains to be evaluated.

Even though some benefits of computer-based decision-support systems have been documented, such systems are slow to be adopted. Moreover, even when computerized guidelines have resulted in demonstrable improvements, often this improvement has been smaller than anticipated. This proposal aims to better understand the barriers to guideline acceptance so that the benefits of computer based decision-support can be realized.

Our organization, Brigham and Women's Hospital, is in a particularly good position to study these issues. We have in place a highly developed clinical information system including an outpatient electronic medical records (EMR) application that has been an active part of the clinical workflow since 1999. The EMR application currently is used by primary care physicians at one of our major medical centers to track their patients' problems, medications, allergies, and health maintenance data. We are developing a new EMR that will be used more broadly across our network, and that features a new interface with added functionality. The new EMR will allow us to evaluate the state of the patient at the time of the visit and generate reminders if the patient is out of compliance for certain guidelines. It also includes outpatient order entry that allows physicians to enter medication and laboratory orders directly into the computer. Decision-support in order entry will allow us to guide physician decision making at the most opportune time, and then evaluate the result of that guidance. For automated decision-support applications to be widely adopted, it is critical that their benefits be demonstrated in a wide variety of situations. We plan to implement several different types of interventions targeted at various phases of the clinical workflow to determine which strategies can achieve the greatest benefit.

Specific Aims:

1. To evaluate the effectiveness of paper-based and interactive computer-based alerts and reminders for improving compliance with guidelines and reducing costs in the ambulatory setting.
2. To evaluate the impact of computer-based tracking and follow-up reminder systems on guideline compliance.
3. To identify and address patient, clinician, and system barriers to the effective use of computer-based clinical decision-support strategies in a diverse array of clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* All physicians in on-site and satellite adult outpatient clinics with the Brigham and Women's Hospital and Massachusetts General Hospital.
* All practices must have adopted our home-grown electronic health record system, the Longitudinal Medical Record, for at least 24 months prior to the start of each intervention trial.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2000-09; Study Completion 2006-12

PRIMARY OUTCOMES:
1) Compliance to guidelines regarding the outpatient laboratory monitoring of prescription medication regiments
2) Compliance to guidelines regarding the follow-up of abnormal test results, including critically abnormal test results, abnormal cholesterol, abnormal HbA1c, abnormal pap smears and abnormal mammogram
3) Compliance to guidelines regarding the management of hypertension in the general ambulatory population and amongst ethnic minority groups
4) Compliance to guidelines regarding the screening and management of osteoporosis

SECONDARY OUTCOMES:
1) Patient satisfaction regarding communication with physicians
2) Physician satisfaction regarding follow-up of abnormal test results

CONTACTS AND LOCATIONS:
Overall Officials: David W Bates, MD MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Poon EG, Haas JS, Louise Puopolo A, Gandhi TK, Burdick E, Bates DW, Brennan TA. Communication factors in the follow-up of abnormal mammograms. J Gen Intern Med. 2004 Apr;19(4):316-23. doi: 10.1111/j.1525-1497.2004.30357.x. PMID 15061740
- [Result] Hickner JM, Fernald DH, Harris DM, Poon EG, Elder NC, Mold JW. Issues and initiatives in the testing process in primary care physician offices. Jt Comm J Qual Patient Saf. 2005 Feb;31(2):81-9. doi: 10.1016/s1553-7250(05)31012-9. PMID 15791767
- [Result] Poon EG, Gandhi TK, Sequist TD, Murff HJ, Karson AS, Bates DW. "I wish I had seen this test result earlier!": Dissatisfaction with test result management systems in primary care. Arch Intern Med. 2004 Nov 8;164(20):2223-8. doi: 10.1001/archinte.164.20.2223. PMID 15534158
- [Result] Poon EG, Wald J, Bates DW, Middleton B, Kuperman GJ, Gandhi TK. Supporting patient care beyond the clinical encounter: three informatics innovations from partners health care. AMIA Annu Symp Proc. 2003;2003:1072. PMID 14728575
- [Result] Gandhi TK, Sequist TD, Poon EG, Karson AS, Murff H, Fairchild DG, Kuperman GJ, Bates DW. Primary care clinician attitudes towards electronic clinical reminders and clinical practice guidelines. AMIA Annu Symp Proc. 2003;2003:848. PMID 14728353
- [Result] Poon EG, Wang SJ, Gandhi TK, Bates DW, Kuperman GJ. Design and implementation of a comprehensive outpatient Results Manager. J Biomed Inform. 2003 Feb-Apr;36(1-2):80-91. doi: 10.1016/s1532-0464(03)00061-3. PMID 14552849
- [Result] Murff HJ, Gandhi TK, Karson AK, Mort EA, Poon EG, Wang SJ, Fairchild DG, Bates DW. Primary care physician attitudes concerning follow-up of abnormal test results and ambulatory decision support systems. Int J Med Inform. 2003 Sep;71(2-3):137-49. doi: 10.1016/s1386-5056(03)00133-3. PMID 14519406
- [Result] Sequist TD, Gandhi TK, Karson AS, Fiskio JM, Bugbee D, Sperling M, Cook EF, Orav EJ, Fairchild DG, Bates DW. A randomized trial of electronic clinical reminders to improve quality of care for diabetes and coronary artery disease. J Am Med Inform Assoc. 2005 Jul-Aug;12(4):431-7. doi: 10.1197/jamia.M1788. Epub 2005 Mar 31. PMID 15802479
- [Derived] Matheny ME, Gandhi TK, Orav EJ, Ladak-Merchant Z, Bates DW, Kuperman GJ, Poon EG. Impact of an automated test results management system on patients' satisfaction about test result communication. Arch Intern Med. 2007 Nov 12;167(20):2233-9. doi: 10.1001/archinte.167.20.2233. PMID 17998497